CLINICAL TRIAL: NCT01543841
Title: A Laboratory Evaluation of Tie-2 Expressing Monocytes (TEMs) in Healthy Volunteers and Patients With Advanced Cancer
Brief Title: Laboratory Testing for Tie-2 Expressing Monocytes (TEMs) in Blood
Status: Completed | Type: Observational
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Other Study IDs: TEMs-DC-001
Record Dates: First submitted 2012-01-19; First posted 2012-03-05 (Estimated); Last update posted 2019-02-15 (Actual); Status verified 2019-02

CONDITIONS: Advanced Cancer; Healthy
Keywords: advanced cancer; healthy; blood sample; TEM; TIE-2 expressing monocytes; ANG1; ANG2

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: None Retained — One tube of whole blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Advanced Cancer: Patients with histologically confirmed metastatic or unresectable solid tumors will have one tube of whole blood (~6mL) collected at the time of venipuncture for routine sample collection. The sample will undergo in vitro stimulation of TEMs with ANG 1 and 3 in the presence or absence of pharmalogic inhibitors, and flow cytometry analysis.
- Healthy Volunteers: Eligible volunteers will have one tube of whole blood (~6mL) collected. The sample will undergo in vitro stimulation of TEMs with ANG 1 and 3 in the presence or absence of pharmalogic inhibitors, and flow cytometry analysis.

SUMMARY:
Tie-2 expressing monocytes (TEMs) are a specific type of blood cell that are present in healthy individuals and in people with cancer. These cells may play a role in the growth of blood vessels (veins/arteries), and may be particularly important in the growth of blood vessels that supply tumours. Understanding how these cells work may therefore help researchers to develop cancer treatments that starve tumors of their blood supply.

This research study involves an analysis of the behaviour of blood cells in response to different drugs in a test tube. The goal is to develop tests that can then be used to monitor patients treated with drugs that target blood vessel growth.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers

  * Ability to understand and the willingness to sign a written informed consent document.
* Patients with advancer cancer

  * Participants must have histologically confirmed metastatic or unresectable solid tumors.
  * Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Healthy volunteers

  * History of cancer within the past 5 years
  * Major medical condition undergoing active therapy
* Patients with advancer cancer

  * Active hematologic malignancy (leukemia, lymphoma, myeloproliferative disorder).
  * Active treatment on a Phase I clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with advanced cancer attending the Phase I clinic and healthy staff at the Princess Margaret Hospital
Sampling Method: Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2012-08; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Characterize the in vitro response of circulating myeloid cells to angiopoeitins-1 and 2 (ANG1 and 2) in the presence or absence of pharmacologic inhibitors | 1 year
  This is an observational correlative laboratory protocol in which one tube of blood from healthy volunteers and cancer patients will be collected to perform in vitro stimulation of TEMs with ANG1 and 2 and flow cytometry analysis, which could serve as a biomarker for future ANG directed therapies. The results of this study will contribute to an improved understanding of ANG-TIE2 signaling in TEMs. Furthermore, this study will contribute directly to the development and optimization of protocols that will be applied a separate Phase I NCI trial of AMG 386 and temsirolimus.

SECONDARY OUTCOMES:
Develop and optimize flow cytometry analyses | 1 year
  This will comprise correlative studies in a separate upcoming Phase I clinical trial.

CONTACTS AND LOCATIONS:
Overall Officials: Lillian Siu, MD, Principal Investigator — Princess Margaret Hospital, Canada
Locations (1):
- Princess Margaret Hospital, Toronto, Ontario, Canada